CLINICAL TRIAL: NCT00081315
Title: Phase II, Randomized, Double-Blind, Multicenter Trial of Subcutaneous Amifostine (Ethyol®) Versus Placebo in the Prevention of Radiochemotherapy-Induced Esophagitis and Pneumonitis in Patients With Unresectable Non-Small Cell Lung Cancer
Brief Title: Subcutaneous Amifostine (Ethyol®) in the Prevention of Radiochemotherapy-Induced Esophagitis and Pneumonitis in Patients With Unresectable Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: MI-CP079
Record Dates: First submitted 2004-04-07; First posted 2004-04-09 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Esophagitis; Pneumonitis; Non-Small Cell Lung Carcinoma
Keywords: - Non-Small cell lung cancer
MeSH Terms: conditions — Esophagitis; Pneumonia; Carcinoma, Non-Small-Cell Lung | interventions — Amifostine

INTERVENTIONS:
Drug: Amifostine

SUMMARY:
The primary objective of this study is to assess the activity of subcutaneous (SC) amifostine on the incidence and severity of acute radiochemotherapy-induced esophagitis in patients with unresectable Stage IIIA or IIIB non-small cell lung cancer (NSCLC) receiving combined modality therapy.

ELIGIBILITY:
You may be eligible for this study if you are 18 years of age or older and:

* Have UnResectable Stage IIIA or IIIB Non Small Cell Lung Cancer
* Have never had prior chemotherapy with Paclitaxel or Carboplatin
* Have never had prior thoracic radiation therapy (XRT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2003-11; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
- Acute radiochemotherapy-induced esophagitis will be assessed from the time of randomization through up to 3 months after completion of radiochemotherapy treatment.

SECONDARY OUTCOMES:
- Acute radiochemotherapy-induced pneumonitis will be assessed until 6 months after the last dose of XRT.

CONTACTS AND LOCATIONS:
Overall Officials: Luz Hammershaimb, M.D., Principal Investigator — MedImmune LLC
Locations (24):
- United States (24):
  - Cedars Sanai, Los Angeles, California
  - Radiation Oncology Center, Sacramento, California
  - The Center for Cancer Care, Torrington, Connecticut
  - Florida Wellcare Alliance, Inverness, Florida
  - Florida Community Cancer Center, New Port Richey, Florida
  - Ormand Memorial Cancer Center, Ormand Beach, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University Community Hospital-Center for Cancer Care, Tampa, Florida
  - University of Kentucky, Lexington, Kentucky
  - St. Agnes Health Care, Baltimore, Maryland
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - Chesapeake Oncology-Hematology Associates, Glen Burnie, Maryland
  - St. John's Medical Research, Springfield, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Beth Israel Hospital, New York, New York
  - Upstate NY Cancer R&E Foundation, Rochester, New York
  - New Hanover Radiation, Wilmington, North Carolina
  - Cancer Center of Upper Delaware Valley, Milford, Pennsylvania
  - Montgomery Cancer Center, Norristown, Pennsylvania
  - Charleston Cancer Center, Charleston, South Carolina
  - The Center for Radiation Oncology, Danville, Virginia
  - Providence Everett Medical Center, Everett, Washington
  - Valley Medical Center, Renton, Washington